CLINICAL TRIAL: NCT05248009
Title: Feasibility of Semi-Permanent Tattoo for Treatment Alignment in Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Ephemeral Solutions Inc. (Industry)
Responsible Party: Principal Investigator, Farzan Siddiqui, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: tattoo_schaff2021
Record Dates: First submitted 2021-09-13; First posted 2022-02-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Tattoo; Pigmentation; Cancer, Treatment-Related
Keywords: radiation therapy; simulation tattoo; cancer; semi-permanent ink
MeSH Terms: conditions — Neoplasms, Second Primary; Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Arm Pilot Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-Permanent Tattoo Ink (Experimental): Semi-Permanent Tattoo Ink
  Interventions: Device: Semi-Permanent Tattoo Ink

INTERVENTIONS:
Device: Semi-Permanent Tattoo Ink — Subjects will receive semi-permanent tattoo ink in place of the permanent ink utilized in the standard of care. Subjects will be monitored during their treatment course and for 15 months following treatment completion.

SUMMARY:
Consenting subjects will receive a semi-permanent tattoo in place of the standard of care permanent tattoo for radiation marking at the time of the radiation planning scan. Subjects will be monitored to ensure alignment is the same with the semi-permanent tattoo as the current standard of care. Subjects will be monitored to ensure there are no skin reactions or other side effects. Subjects will be followed for 15 months and will send pictures to the treatment team to ensure that the tattoo fades away within 12 months as expected.

DETAILED DESCRIPTION:
Over 3 million patients are treated each year with radiation therapy, with most of these patients receiving permanent tattoos for treatment alignment. The purpose of these tattoos is to ensure accurate initial patient position prior to treatment. In the case where further on-board imaging such as x-ray or cone-beam CT is used, the radiation tattoos help minimize large shifts which increase treatment time and radiation exposure as further imaging may be required. The tattoos are simple and effective, but also permanent. These permanent tattoos serve as a daily reminder of prior radiation therapy in cancer survivors which may have a negative psychological impact on the patients quality of life. Due to this, many patients will seek laser tattoo removal after completing radiation therapy. There have been attempts at non-permanent tattoo options such as henna as well as omitting tattoos altogether using surface imaging. Unfortunately, henna and other temporary tattoos start to fade quickly and do not last the 6-8 weeks required for longer radiation courses. This means that the tattoos must be reapplied over the course of treatment which can introduce inaccuracies as well as prolongs the treatment time.

A novel semi-permanent ink has been developed and recently released which begins to fade after 6 months and disappears after about 1 year. This is the first ink of its kind and is delivered using a needle into the dermis just like a permanent tattoo, however it is able to be resorbed by the body after approximately 1 year. While the original purpose is for cosmetic tattoos it has a possible application in medical tattoos for radiation therapy.

It is the goal of this study to show that the semi-permanent ink is safe, allows for accurate alignment of the patient prior to treatment, lasts long enough for a full treatment course, and fades over time. The goal in subsequent studies is to improve patient quality of life by decreasing the negative psychological impact of having permanent tattoos following radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring medical tattoo for treatment alignment.
* Patient being treated with some form of image guidance including kV, MV, or cone-beam CT.
* Age ≥ 18.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients will engage in the informed consent process and provide study-specific informed consent prior to study entry and must be willing to have photos taken of their tattoos through the treatment and follow-up process and may be required to take pictures of their own tattoo to submit to the research team.
* Patient able to send picture of tattoo via secure messaging.

Exclusion Criteria:

* Known allergies or hypersensitivity to tattoo ink.
* Personal or religious objection to medical tattooing.
* Autoimmune or skin disorders which may be worsened by medical tattooing.
* Inability to complete the required forms; however, verbal completion is adequate if recorded on the consent documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Skin Adverse Events - During Treatment | Subjects will be followed weekly during their treatment course
  Adverse events related to the tattooing process including skin toxicity during the completion of radiation therapy will be assessed using Common Terminology Criteria for Adverse Events (CTCAE v5). The type, incidence, severity, timing, serious, and relatedness of AE and laboratory abnormalities will be reported and tabulated. The CTCAE is assessed according to grades 1-5, where grade 5 constitutes the highest severity and worse outcome.

SECONDARY OUTCOMES:
Mean 3D Vector Shifts | Subjects will be followed until completion of their 5-7 week treatment course
  The primary endpoint is the mean 3D vector shifts as determined by couch shifts from initial setup using tattoo to final treatment position which is verified and shifted based on further imaging including x-ray or cone-beam CT scan. Mean and standard deviation of 3D vector shifts will be summarized, and t-test or Mann-Whitney test will be used to compared with historical data.
Skin Adverse Events - Post Treatment | Subjects will be followed every 3 months for 15 months after completion of treatment
  Adverse events related to the tattooing process including skin toxicity during the completion of radiation therapy will be assessed using Common Terminology Criteria for Adverse Events (CTCAE v5). The type, incidence, severity, timing, serious, and relatedness of AE and laboratory abnormalities will be reported and tabulated. The CTCAE is assessed according to grades 1-5, where grade 5 constitutes the highest severity and worse outcome.
Change from Baseline Tattoo Visibility at 15 Months | Subjects will be followed weekly during their 5-7 week treatment course and every 3 months for 15 months after completion of treatment
  The second primary endpoint will be tattoo visibility which will be scored on a 4-point scale and assessed until end of follow up. The scoring ranges from 0-3, with 0 representing not visible and 3 representing easily visible. This will be assessed weekly during treatment by both the treating physician/research team as well as the patient. Tattoo fading will be compared to baseline which is measured during the first week of radiation therapy to give time to heal after tattoo placement at time of simulation. Tattoo visibility score from baseline for each patient will be summarized by spaghetti plot. Time to complete invisible will be summarized by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Farzan Siddiqui, MD PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryant AK, Banegas MP, Martinez ME, Mell LK, Murphy JD. Trends in Radiation Therapy among Cancer Survivors in the United States, 2000-2030. Cancer Epidemiol Biomarkers Prev. 2017 Jun;26(6):963-970. doi: 10.1158/1055-9965.EPI-16-1023. Epub 2017 Jan 17. PMID 28096199
- [Background] Bregnhoj A, Haedersdal M. Q-switched YAG laser vs. punch biopsy excision for iatrogenic radiation tattoo markers--a randomized controlled trial. J Eur Acad Dermatol Venereol. 2010 Oct;24(10):1183-6. doi: 10.1111/j.1468-3083.2010.03617.x. PMID 20236380
- [Background] Wurstbauer K, Sedlmayer F, Kogelnik HD. Skin markings in external radiotherapy by temporary tattooing with henna: improvement of accuracy and increased patient comfort. Int J Radiat Oncol Biol Phys. 2001 May 1;50(1):179-81. doi: 10.1016/s0360-3016(01)01439-0. PMID 11316562
- [Background] Jimenez RB, Batin E, Giantsoudi D, Hazeltine W, Bertolino K, Ho AY, MacDonald SM, Taghian AG, Gierga DP. Tattoo free setup for partial breast irradiation: A feasibility study. J Appl Clin Med Phys. 2019 Apr;20(4):45-50. doi: 10.1002/acm2.12557. PMID 30945803